CLINICAL TRIAL: NCT01720524
Title: A MULTI-CENTRE, RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE-BLIND, TWO-ARMED, PARALLEL GROUP STUDY TO EVALUATE EFFICACY AND SAFETY OF IV SILDENAFIL IN THE TREATMENT OF NEONATES WITH PERSISTENT PULMONARY HYPERTENSION OF THE NEWBORN (PPHN) OR HYPOXIC RESPIRATORY FAILURE AND AT RISK FOR PPHN, WITH A LONG TERM FOLLOW-UP INVESTIGATION OF DEVELOPMENTAL PROGRESS 12 AND 24 MONTHS AFTER COMPLETION OF STUDY TREATMENT
Brief Title: A Study To Evaluate Safety And Efficacy Of IV Sildenafil In The Treatment Of Neonates With Persistent Pulmonary Hypertension Of The Newborn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481316; 2012-002619-24 (EudraCT Number)
Record Dates: First submitted 2012-09-17; First posted 2012-11-02 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Hypertension, Familial Persistent, of the Newborn
Keywords: persistent pulmonary hypertension; newborn; neonates; iv sildenafil; hypoxic respiratory failure and at risk of persistent pulmonary hypertension of the newborn
MeSH Terms: conditions — Persistent Fetal Circulation Syndrome | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): iv placebo of normal saline or 10% dextrose
  Interventions: Drug: placebo
- sildenafil (Experimental): Active study drug
  Interventions: Drug: iv sildenafil

INTERVENTIONS:
Drug: placebo — IV placebo or 0.9% sodium chloride or 10% dextrose. Infusion rate based on weight.
  Arms: placebo
Drug: iv sildenafil — loading dose of 0.1 mg/kg over 30 minutes followed by maintenance dose of 0.03 mg/kg/h. To infuse minimum 48 hours and maximum of 14 days.
  Other Names: revatio
  Arms: sildenafil

SUMMARY:
This study will evaluate whether IV sildenafil can reduce the time on inhaled nitric oxide treatment and reduce the failure rate of available treatments for persistent pulmonary hypertension of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with persistent pulmonary hypertension of the newborn
* Age <=96 hours and >=34 weeks gestational age
* Oxygenation Index >15 and <60
* Concurrent treatment with inhaled nitric oxide and >=50% oxygen

Exclusion Criteria:

* Prior or immediate need for extracorporeal membrane oxygenation or cardiopulmonary resuscitation
* Expected duration of mechanical ventilation <48 hours
* Profound hypoxemia
* Life-threatening or lethal congenital anomaly

Ages: 0 Days to 4 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2013-08-05 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (19):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California Davis Medical Center, Sacramento, California
  - University of California Davis, Sacramento, California
  - Children´s National Medical Center, Washington D.C., District of Columbia
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Sydney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OU Follow-Up Program, PREMIEr Clinic, Children's Hospital, Oklahoma City, Oklahoma
  - OU Neonatal Intensive Care Unit at Children's Hospital, Oklahoma City, Oklahoma
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Henry Zarrow Neonatal Intensive Care Unit, Children's Hospital at Saint Francis, Tulsa, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Seattle Children's Research Institute, Seattle, Washington
  - Seattle Childrens Hospital, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
- CHUL du CHU de Quebec, Québec, Quebec, Canada
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Neonatalklinikken Rigshospitalet, 5024, Copenhagen Ø
- France (5):
  - Centre Hospitalier et Regional de Lille - Hopital Jeanne de Flandre, Lille
  - Centre Hospitalier et Régional de Lille,, Lille
  - Hôpital de la Conception Assistance Publique-Hôpitaux de Marseille, Marseille
  - CHU Robert Debré, Paris
  - Hopital NECKER - Enfants Malades, Paris
- University Hospital of Leipzig, Leipzig, Germany
- Neonatologia Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
- Netherlands (2):
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus MC, Sophia Children's hospital, Rotterdam
- Haukeland University Hospital, Bergen, Haukeland, Norway
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona / Spain
  - Hospital General Universitario Gregorio Marañon, Madrid
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (4):
  - St. Michael's Hospital, Bristol
  - Leicester Royal Infirmary, Leicester
  - Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester
  - Great Ormond Street Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Pierce CM, Zhang MH, Jonsson B, Iorga D, Cheruvu N, Balagtas CC, Steinhorn RH. Efficacy and Safety of IV Sildenafil in the Treatment of Newborn Infants with, or at Risk of, Persistent Pulmonary Hypertension of the Newborn (PPHN): A Multicenter, Randomized, Placebo-Controlled Trial. J Pediatr. 2021 Oct;237:154-161.e3. doi: 10.1016/j.jpeds.2021.05.051. Epub 2021 May 27. PMID 34052232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481316&StudyName=A%20Study%20To%20Evaluate%20Safety%20And%20Efficacy%20Of%20IV%20Sildenafil%20In%20The%20Treatment%20Of%20Neonates%20With%20Persistent%20Pulmonary%20Hypertension%20Of%20The%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was planned in two parts Part A (double-blind phase) and Part B (long-term, non-intervention phase).
Pre-assignment Details: Neonates with persistent pulmonary hypertension of the newborn (PPHN) or hypoxic respiratory failure (HRF) and at risk of PPHN who were receiving inhaled nitric oxide (iNO) treatment were evaluated in this study.
Groups:
- IV Sildenafil: Part A: Participants received sildenafil intravenously based on their body weight at a loading dose of 0.1 milligrams per kg (mg/kg) for 30 minutes on Day 1 followed by a maintenance dose of 0.03 milligrams per kg per hour (mg/kg/hr), for a minimum of 2 days and maximum of 14 days. Infusion continuation was upon investigator discretion in view of participants' safety and well-being. Part B: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
- Placebo: Participants received placebo (0.9 % normal saline or dextrose 10%) at a rate matched to sildenafil infusion, intravenously, based on participant's weight, for a minimum of 2 days and maximum of 14 days. Infusion continuation was upon investigator discretion in view of participants' safety and well-being. Part B: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
Period: Part A
Arm/Group | IV Sildenafil | Placebo
Started | 29 | 30
Completed | 22 | 18
Not Completed | 7 | 12
Not completed — Insufficient Clinical Response | 2 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Missed 28 day follow-up visit | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Part B
Arm/Group | IV Sildenafil | Placebo
Started | 27 (Participants who did not complete Part A could also participate in Part B.) | 26 (Participants who did not complete Part A could also participate in Part B.)
Completed | 22 | 17
Not Completed | 5 | 9
Not completed — No longer willing to participate in study | 1 | 4
Not completed — Other | 2 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants treated with study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Sildenafil | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: days] | 1.7 (0.90) | 1.9 (0.75) | 1.8 (0.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 23 | 29 | 52
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 5 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 19 | 16 | 35
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time on Inhaled Nitric Oxide (iNO) Treatment After Initiation of Intravenous (IV) Study Drug For Participants Without Treatment Failure
Description: Time in days, on iNO treatment, for participants without iNO treatment failure, was calculated 14 days from the initiation of IV study drug or hospital discharge, whichever occurred first. iNO treatment failure was defined as need for additional treatment targeting PPHN, need for extra corporeal membrane oxygenation (ECMO), or death during the study.
Time Frame: 14 days from the initiation of IV study drug or hospital discharge, whichever occurs first (maximum of 14 days)
Population: The intent-to-treat population (ITT) included all randomized participants treated with study treatment. Here "Overall number of participants analyzed" signifies number of participants without iNO treatment failure.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 21 | 24
days | 4.1 [2.58 to 5.58] | 4.1 [2.70 to 5.50]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Test type: Superiority; p = 0.9850, ANCOVA; Least square (LS) mean difference = 0.0, 95% CI 2-sided [-2.08 to 2.04], Standard Error of Mean 1.02

2. Primary Outcome: Treatment Failure Rate
Description: Treatment failure rate was defined as percentage of participants who needed additional treatment targeting PPHN, needed ECMO, or died during the study.
Time Frame: 14 days from the initiation of IV study drug or hospital discharge, whichever occurs first (maximum of 14 days)
Population: The ITT population included all randomized participants treated with study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
percentage of participants | 27.6 [11.3 to 43.9] | 20.0 [5.7 to 34.3]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Test type: Superiority; p = 0.4935, Chi-squared; Difference in percentage = 7.6, 95% CI 2-sided [-14.1 to 29.3]

3. Secondary Outcome: Time From Initiation of Intravenous (IV) Study Drug to Final Weaning of Mechanical Ventilation
Description: Time in days, from initiation of IV study drug to final weaning of mechanical ventilation among participants achieving final weaning of mechanical ventilation for PPHN was evaluated. Kaplan-Meier method was used for estimation. For participants with mechanical ventilation beyond 336 hours (14 days) from initiation of IV study drug, data was censored at 14 days.
Time Frame: 14 days from the initiation of IV study drug or hospital discharge, whichever occurs first (maximum of 14 days)
Population: The ITT population included all randomized participants treated with study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
days | 8.3 [5.46 to 11.75] | 7.3 [5.46 to 10.78]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Test type: Superiority; p = 0.9885, Log Rank

4. Secondary Outcome: Time From Initiation of Intravenous (IV) Study Drug to First Treatment Failure
Description: Time in days, from initiation of IV study drug to first treatment failure (defined as need for additional treatment targeting PPHN, need for ECMO, or death) for participants with treatment failure was evaluated. Kaplan-Meier method was used for estimation. For participants without treatment failure by the endpoint assessment date, data was censored at the endpoint assessment date.
Time Frame: 14 days from the initiation of IV study drug or hospital discharge, whichever occurs first (maximum of 14 days)
Population: The ITT population included all randomized participants treated with study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
days | NA [NA to NA] — Due to low number of participants with events, Kaplan-Meier estimates of median, upper and lower limit of CI could not be estimated/calculated. | NA [NA to NA] — Due to low number of participants with events, Kaplan-Meier estimates of median, upper and lower limit of CI could not be estimated/calculated.
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Test type: Superiority; p = 0.4910, Log Rank

5. Secondary Outcome: Percentage of Participants With Individual Components of Treatment Failure
Description: Percentage of participants with individual components of treatment failure (need to start additional treatment targeting PPHN, need to start ECMO, or death) were evaluated. Some participants could have had multiple qualifying events for treatment failure.
Time Frame: 14 days from the initiation of IV study drug or hospital discharge, whichever occurs first (maximum of 14 days)
Population: The ITT population included all randomized participants treated with study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
percentage of participants
  Additional Treatment Targeting PPHN | 13.8 [3.9 to 31.7] | 10.0 [2.1 to 26.5]
  ECMO | 10.3 [2.2 to 27.4] | 10.0 [2.1 to 26.5]
  Death | 6.9 [0.8 to 22.8] | 0.0 [0.0 to 11.6]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Additional Treatment; Test type: Superiority; p = 0.7065, Fisher Exact; Difference in Percentage = 3.8, 95% CI 2-sided [-15.2 to 22.9]
Statistical Analysis 2: Comparison: IV Sildenafil vs Placebo; ECMO; Test type: Superiority; p > 0.999, Fisher Exact; Difference in Percentage = 0.3, 95% CI 2-sided [-18.5 to 18.5]
Statistical Analysis 3: Comparison: IV Sildenafil vs Placebo; Death; Test type: Superiority; p = 0.2373, Fisher Exact; Difference in Percentage = 6.9, 95% CI 2-sided [-5.5 to 22.8]

6. Secondary Outcome: Change From Baseline in Oxygenation Index (OI) at Hours 6, 12 and 24 Post-Infusion
Description: Oxygenation index was calculated as the product of fraction of inspired oxygen (FiO2) and mean airway pressure divided by partial pressure of oxygen dissolved in arterial blood (PaO2) [(FiO2*mean airway pressure)/PaO2] measured in centimeter of water per millimeter of mercury (cmH2O/mmHg). FiO2 is the measure of oxygen concentration that is breathed. Mean airway pressure is defined as an average of the airway pressure throughout the respiratory cycle. PaO2 is the measure of oxygen level dissolved in the arterial blood.
Time Frame: Baseline, Hours 6, 12 and 24 after start of infusion
Population: The ITT population included all randomized participants treated with study treatment. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Least Squares Mean (95% Confidence Interval); unit: cmH2O/mmHg
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
cmH2O/mmHg
  Change at Hour 6: number analyzed (Participants) | 29 | 22
  Change at Hour 6 | -4.2 [-11.64 to 3.34] | -8.0 [-16.63 to 0.57]
  Change at Hour 12: number analyzed (Participants) | 28 | 22
  Change at Hour 12 | -4.1 [-10.51 to 2.23] | -8.2 [-15.42 to -1.04]
  Change at Hour 24: number analyzed (Participants) | 18 | 17
  Change at Hour 24 | -11.6 [-15.40 to -7.83] | -9.5 [-13.36 to -5.57]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Hour 6; Test type: Superiority; p = 0.4984, ANCOVA; LS Mean Difference = 3.9, 95% CI 2-sided [-7.5 to 15.3]
Statistical Analysis 2: Comparison: IV Sildenafil vs Placebo; Hour 12; Test type: Superiority; p = 0.3956, ANCOVA; LS Mean Difference = 4.1, 95% CI 2-sided [-5.5 to 13.7]
Statistical Analysis 3: Comparison: IV Sildenafil vs Placebo; Hour 24; Test type: Superiority; p = 0.4249, ANCOVA; LS Mean Difference = -2.2, 95% CI 2-sided [-7.6 to 3.3]

7. Secondary Outcome: Change From Baseline in Differential Saturation at Hours 6, 12 and 24 Post-Infusion
Description: Differential oxygenation saturation is a simple way to detect the right-to left shunting at ductus arteriosus using 2 pulse oximeters. It is the difference between pre-ductal and post-ductal sites pulse oxygen saturation (SpO2). Where, pre-duct refers to right upper extremity and post-duct refers to lower limb. Oxygenation saturation is measured as percentage of hemoglobin binding sites occupied by oxygen in the blood.
Time Frame: Baseline, Hours 6, 12 and 24 after start of infusion
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of hemoglobin
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
percentage of hemoglobin
  Change at Hour 6: number analyzed (Participants) | 26 | 19
  Change at Hour 6 | 1.5 [-1.79 to 4.80] | 0.8 [-3.10 to 4.62]
  Change at Hour 12: number analyzed (Participants) | 25 | 19
  Change at Hour 12 | -1.2 [-7.65 to 5.21] | 6.7 [-0.65 to 14.12]
  Change at Hour 24: number analyzed (Participants) | 19 | 14
  Change at Hour 24 | 1.2 [-7.15 to 9.49] | 9.3 [-0.40 to 19.08]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Hour 6; Test type: Superiority; p = 0.7686, ANCOVA; LS Mean Difference = 0.7, 95% CI 2-sided [-4.3 to 5.8]
Statistical Analysis 2: Comparison: IV Sildenafil vs Placebo; Hour 12; Test type: Superiority; p = 0.1112, ANCOVA; LS Mean Difference = -8.0, 95% CI 2-sided [-17.8 to 1.9]
Statistical Analysis 3: Comparison: IV Sildenafil vs Placebo; Hour 24; Test type: Superiority; p = 0.2089, ANCOVA; LS Mean Difference = -8.2, 95% CI 2-sided [-21.2 to 4.8]

8. Secondary Outcome: Change From Baseline in Ratio of Partial Pressure of Oxygen in Arterial Blood to Fraction of Inspired Oxygen (P/F) at Hours 6, 12 and 24
Description: The ratio of partial pressure of arterial oxygen to fraction of inspired oxygen is a ratio between the oxygen level in the arterial blood and the oxygen concentration that is breathed. It helps to determine the degree of any problems with how the lungs transfer oxygen to the blood.
Time Frame: Baseline, Hours 6, 12 and 24 after start of infusion
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
ratio
  Change at Hour 6: number analyzed (Participants) | 29 | 23
  Change at Hour 6 | 45.3 [17.21 to 73.37] | 8.1 [-23.48 to 39.60]
  Change at Hour 12: number analyzed (Participants) | 28 | 24
  Change at Hour 12 | 43.4 [16.76 to 70.13] | 16.9 [-11.97 to 45.68]
  Change at Hour 24: number analyzed (Participants) | 20 | 17
  Change at Hour 24 | 94.6 [18.52 to 170.69] | 14.7 [-67.83 to 97.25]
Statistical Analysis 1: Comparison: IV Sildenafil vs Placebo; Hour 6; Test type: Superiority; p = 0.0829, ANCOVA; LS Mean Difference = 37.2, 95% CI 2-sided [-5.0 to 79.5]
Statistical Analysis 2: Comparison: IV Sildenafil vs Placebo; Hour 12; Test type: Superiority; p = 0.1802, ANCOVA; LS Mean Difference = 26.6, 95% CI 2-sided [-12.7 to 65.9]
Statistical Analysis 3: Comparison: IV Sildenafil vs Placebo; Hour 24; Test type: Superiority; p = 0.1576, ANCOVA; LS Mean Difference = 79.9, 95% CI 2-sided [-32.5 to 192.2]

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Sildenafil and Its Metabolite
Description: Cmax was obtained for Sildenafil and its major metabolite UK-103,320.
Time Frame: Loading dose, Day 1: prior to the start of infusion, 5, 30 minutes after end of loading infusion; Maintenance dose: 48 to 72, 96 to 120 hours during infusion and immediately prior to end of maintenance infusion (up to maximum on Day 14)
Population: Pharmacokinetic (PK) analysis set included all participants randomized and treated who had at least 1 concentration during whole treatment period.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | IV Sildenafil
Number analyzed (Participants) | 25
nanogram per milliliter
  Loading dose: Sildenafil | 52.64 (27.91)
  Loading dose: UK-103320 | 1.04 (1.68)
  Maintenance dose: Sildenafil | 78.12 (48.63)
  Maintenance dose: UK-103320 | 21.65 (11.57)

10. Secondary Outcome: Total Plasma Clearance (CL) of Sildenafil and Its Metabolite
Description: CL is volume of the body fluid/ plasma from which the drug or the metabolite is completely removed per unit time. CL was obtained for Sildenafil and its major metabolite UK-103,320.
Time Frame: Loading dose: prior to the start of infusion, 5, 30 minutes after end of loading infusion on Day 1; Maintenance dose: between 48 to 72, 96 to 120 hours during infusion and immediately prior to end of infusion on Day 1
Population: PK analysis set included all participants randomized and treated who had at least 1 concentration during whole treatment period.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | IV Sildenafil
Number analyzed (Participants) | 25
Liters/hour
  Sildenafil | 1.78 (0.89)
  UK-103,320 | 5.05 (2.25)

11. Secondary Outcome: Central Volume of Distribution (Vc) of Sildenafil and Its Metabolite
Description: Vc is the hypothetical volume into which a drug or a metabolite initially distributes upon administration. It was determined by using a population-based analysis, non-linear mixed-effects modeling (NONMEM), version 7.4.0. Vc was calculated for Sildenafil and its major metabolite, UK-103,320.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | IV Sildenafil
Number analyzed (Participants) | 25
Liters
  Sildenafil | 8.76 (1.8)
  UK-103,320 | 15.96 (11.20)

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent are events between first infusion of study drug and up to 31 days after end of study drug infusion (up to 45 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 31 days after end of study drug infusion (up to 45 days)
Population: The safety population included all participants treated with study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
Participants
  AEs | 22 | 19
  SAEs | 7 | 2

13. Secondary Outcome: Number of Treatment-Emergent Adverse Events (AEs) According to Severity
Description: AE: untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE: AE resulting in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent are events between first infusion of study drug and up to 31 days after end of study drug infusion (up to 45 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs. Severity criteria: mild=did not interfere with subject's usual function; moderate=interfered to some extent with participant's usual function and severe=interfered significantly with participant's usual function. Missing baseline severities were imputed as mild.
Time Frame: Baseline up to 31 days after end of study drug infusion (up to 45 days)
Population: The safety population included all participants treated with study treatment.
Measure: Number; unit: events
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 30
events
  Mild | 49 | 42
  Moderate | 29 | 24
  Severe | 12 | 17

14. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria for laboratory values: Hematology: hemoglobin, hematocrit, red blood cell count <0.8*lower limit of normal (LLN), platelets<0.5*LLN, >1.75*upper limit of normal (ULN), white blood cells count <0.6*LLN, >1.5*ULN; Liver function: total and direct bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN, total protein <0.8*LLN, >1.2*ULN; Renal function: blood urea nitrogen, creatinine >1.3*ULN; Electrolytes: sodium <0.95*LLN, >1.05*ULN, potassium, chloride, calcium, bicarbonate (venous) <0.9*LLN, >1.1*ULN.
Time Frame: Up to 14 days from initiation of study drug infusion
Population: The safety population included all participants treated with study treatment. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 29 | 28
Participants | 27 | 22

15. Secondary Outcome: Part B: Composite Scores of Cognitive, Language, and Motor Developmental Progress of Participants as Assessed by Bayley Scales of Infant and Toddler Development Third Edition (Bayley-III)
Description: Bayley-III assesses infant and toddler development across five domains: cognitive, language, motor, social-emotional (SE), and adaptive behavior (AB). Assessments of the cognitive, language, and motor domains conducted using items administered to the child; assessments of the SE and AB domains conducted using the primary caregiver's responses to a questionnaire. Score ranges: cognitive scale 0-91, language scale 0-97 and motor scale 0-132, where higher scores indicated better cognitive function, communication and motor skills respectively. Raw scores of cognitive, language and motor domains were converted to composite scores. Composite scores of cognitive, language and motor developmental scales ranged from a scale of 40 to 160, where higher score indicated stronger skills and abilities. In this outcome measure composite scores for infants and toddlers were reported at month 12 and 24.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: Part B safety analysis set included all participants enrolled in Part B of the study for data analyses on developmental progress, audiological, neurological and ophthalmological assessment, and safety. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 19 | 13
units on a scale
  Cognitive Development: Month 12: number analyzed (Participants) | 19 | 12
  Cognitive Development: Month 12 | 97.5 (16.14) | 94.5 (14.18)
  Cognitive Development: Month 24: number analyzed (Participants) | 17 | 13
  Cognitive Development: Month 24 | 97.4 (18.12) | 97.3 (14.95)
  Language Development: Month 12: number analyzed (Participants) | 18 | 12
  Language Development: Month 12 | 99.5 (16.86) | 94.7 (10.25)
  Language Development: Month 24: number analyzed (Participants) | 16 | 11
  Language Development: Month 24 | 96.7 (21.91) | 95.8 (17.70)
  Motor Development: Month 12: number analyzed (Participants) | 19 | 12
  Motor Development: Month 12 | 93.1 (16.10) | 88.2 (14.61)
  Motor Development: Month 24: number analyzed (Participants) | 17 | 12
  Motor Development: Month 24 | 99.0 (19.59) | 105.3 (24.00)

16. Secondary Outcome: Part B: Composite Scores of Social-Emotional and Adaptive Behavior Questionnaire as Assessed by Bayley Scales of Infant and Toddler Development Third Edition (Bayley-III)
Description: The Bayley-III assesses infant and toddler development across five domains: cognitive, language, motor, social-emotional (SE), and adaptive behavior (AB). Assessments of the cognitive, language, and motor domains conducted using items administered to the child; assessments of the SE and AB domains conducted using the primary caregiver's responses to a questionnaire. The questionnaire comprises the SE scale (35 items) and the AB scale (241 items). Raw scores of SE and AB were converted to composite scores. Composite scores for SE and AB scale ranged from 40 to 160, where higher scores indicated better social-emotional skills and adaptive behavior in child. In this outcome measure composite scores for parent/caregiver were reported at month 24.
Time Frame: Month 24 after end of study treatment in Part A (Day 1 to 14)
Population: Part B safety analysis set included all participants enrolled in Part B of the study for data analyses on developmental progress, audiological, neurological and ophthalmological assessment, and safety. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 15 | 8
units on a scale
  Social-Emotional Development | 104.5 (21.40) | 112.5 (18.13)
  Adaptive Behavior Development | 91.6 (15.66) | 98.3 (12.44)

17. Secondary Outcome: Part B: Number of Participants With Eye Movement Disorders as Assessed by Eye Examination
Description: Standard age-appropriate ophthalmological examinations were used to assess eye movement disorders (presence of amblyopia, strabismus, and nystagmus) at month 12 and 24. In this outcome measure, data have been reported for right and left eye separately. Rows according to eye movement disorder categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 16 | 14
Participants
  Strabismus Present, Right Eye: Month 12 | 0 | 1
  Strabismus Present, Left Eye: Month 12 | 0 | 1
  Strabismus Present, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  Strabismus Present, Right Eye: Month 24 | 1 | 0
  Strabismus Present, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  Strabismus Present, Left Eye: Month 24 | 1 | 0
  Nystagmus Present, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  Nystagmus Present, Left Eye: Month 24 | 0 | 1

18. Secondary Outcome: Part B: Visual Acuity of Verbal Participants as Assessed by Ophthalmological Assessment
Description: Standard age-appropriate ophthalmological examinations were used to assess visual acuity (performed differently for children able of verbal interaction) through visual acuity chart (VAC) quantitative, counting finger (CF), hand motion (HM), light perception (LP), no light perception (NLP) and missing at month 12 and 24. In this outcome measure, data have been reported for right and left eye separately. Rows according to visual acuity categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 16 | 14
Participants
  VAC Quantitative, Right Eye: Month 12 | 2 | 1
  HM, Right Eye: Month 12 | 0 | 2
  LP, Right Eye: Month 12 | 1 | 0
  Missing, Right Eye: Month 12 | 13 | 11
  VAC Quantitative, Left Eye: Month 12 | 2 | 1
  HM, Left Eye: Month 12 | 0 | 2
  LP, Left Eye: Month 12 | 1 | 0
  Missing, Left Eye: Month 12 | 13 | 11
  VAC Quantitative, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  VAC Quantitative, Right Eye: Month 24 | 6 | 5
  HM, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  HM, Right Eye: Month 24 | 1 | 0
  Missing, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  Missing, Right Eye: Month 24 | 5 | 7
  VAC Quantitative, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  VAC Quantitative, Left Eye: Month 24 | 6 | 5
  Missing, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  Missing, Left Eye: Month 24 | 6 | 7

19. Secondary Outcome: Part B: Visual Acuity of Non-Verbal Participants as Assessed by Ophthalmological Assessment
Description: Standard age-appropriate ophthalmological examinations were used to assess visual acuity (performed differently for children unable of verbal interaction) through fixates and follows (included central, steady and maintained), light perception (wince to light), no light perception, and missing at month 12 and 24. In this outcome measure, data have been reported for right and left eye separately. Rows according to visual acuity categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 16 | 14
Participants
  Fixates and Follows, Right Eye: Month 12 | 15 | 13
  Light Perception, Right Eye: Month 12 | 0 | 1
  Missing, Right Eye: Month 12 | 1 | 0
  Fixates and Follows, Left Eye: Month 12 | 15 | 13
  Light Perception, Left Eye: Month 12 | 0 | 1
  Missing, Left Eye: Month 12 | 1 | 0
  Fixates and Follows, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  Fixates and Follows, Right Eye: Month 24 | 5 | 9
  Missing, Right Eye: Month 24: number analyzed (Participants) | 12 | 12
  Missing, Right Eye: Month 24 | 7 | 3
  Fixates and Follows, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  Fixates and Follows, Left Eye: Month 24 | 5 | 9
  Missing, Left Eye: Month 24: number analyzed (Participants) | 12 | 12
  Missing, Left Eye: Month 24 | 7 | 3

20. Secondary Outcome: Part B: Visual Acuity of Verbal Participants as Assessed by LogMAR Through Visual Acuity Chart
Description: Standard age-appropriate ophthalmological examinations were used to assess visual acuity (performed differently for children able of verbal interaction) at month 12 and 24. Visual acuity (VA) of verbal children was assessed for each eye using the Snellen method, where logarithm of minimum angle of resolution (logMAR) units were derived from the Snellen ratios. Participants had to read letters from the chart at a distance of 20 feet/6 meter or 4 meter. VA (Snellen ratio) = distance between the chart and participant, divided by distance at which participant was able to see/read chart without impairment; expressed as decimal, logMAR = log10 (1/decimal VA). In this outcome measure, data have been reported for right and left eye separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 6 | 6
LogMAR
  Right Eye: Month 12: number analyzed (Participants) | 6 | 3
  Right Eye: Month 12 | 0.45 (0.394) | 0.57 (0.513)
  Left Eye: Month 12: number analyzed (Participants) | 6 | 3
  Left Eye: Month 12 | 0.47 (0.372) | 0.57 (0.513)
  Right Eye: Month 24: number analyzed (Participants) | 6 | 4
  Right Eye: Month 24 | 0.20 (0.155) | 0.28 (0.299)
  Left Eye: Month 24 | 0.20 (0.155) | 0.35 (0.409)

21. Secondary Outcome: Part B: Visual Status of Participants With Abnormality as Assessed by Eye Examination of the Anterior and Posterior Segments
Description: Standard age-appropriate ophthalmological examinations were used to assess examination of anterior and posterior chamber for abnormality in lids, conjunctiva, cornea, anterior chamber, lens, iris, pupil, extraocular muscle movement and eye movements at month 12 and 24. In this outcome measure, data have been reported for right and left eye separately. Rows according to visual status categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 17 | 15
Participants
  Anterior Segment (Lids), Right Eye: Month 12 | 0 | 1
  Anterior Segment (Lids), Left Eye: Month 12 | 0 | 1
  Anterior Segment (Extraocular muscle movements), Right Eye: Month 24: number analyzed (Participants) | 13 | 11
  Anterior Segment (Extraocular muscle movements), Right Eye: Month 24 | 1 | 0
  Anterior Segment (Extraocular muscle movements), Left Eye: Month 24: number analyzed (Participants) | 13 | 11
  Anterior Segment (Extraocular muscle movements), Left Eye: Month 24 | 1 | 0

22. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Behavior Hearing Assessment Through Pure Tone Audiometry Test
Description: Audiological evaluations of participants were recorded and reported using behavior hearing assessment through pure tone audiometry test which includes participants with normal, abnormal, incomplete/inconclusive behavior at month 12 and 24.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 16 | 12
Participants
  Normal Behavioral Assessment: Month 12 | 11 | 8
  Abnormal Behavioral Assessment: Month 12 | 1 | 4
  Incomplete/Inconclusive Behavioral Assessment: Month 12 | 4 | 0
  Normal Behavioral Assessment: Month 24 | 13 | 8
  Abnormal Behavioral Assessment: Month 24 | 0 | 2
  Incomplete/Inconclusive Behavioral Assessment: Month 24 | 3 | 2

23. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Bone Conduction Through Pure Tone Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by bone conduction assessment through pure tone audiometry test which included participants with sensorineural hearing loss, conductive hearing loss, mixed hearing loss, neural, and unspecified at month 12 and 24. Rows according to bone conduction categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 1 | 2
Participants
  Conductive Hearing Loss: Month 12 | 0 | 1
  Unspecified: Month 12 | 1 | 1
  Conductive Hearing Loss: Month 24: number analyzed (Participants) | 0 | 1
  Conductive Hearing Loss: Month 24 |  | 1

24. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Air Conduction Via Phones/Headphones Through Pure Tone Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by air conduction via phones/headphones through pure tone audiometry test which included participants with hearing loss ranged from less than or equal to (<=) 20 decibel hearing loss (DB HL), 21-40 DB HL, 41-70 DB HL, 71-90 DB HL, greater than (>) 90 DB HL or no response, and missing at frequencies ranged from 500 Hertz (Hz) to 8000 Hz at month 12 and 24. In this outcome measure, data have been reported for right and left ear separately. Rows according to air conduction categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 8 | 5
Participants
  Right Ear, 500 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 500 Hz, <=20 DB HL: Month 12 | 3 | 4
  Right Ear, 500 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 500 Hz, 21 - 40 DB HL: Month 12 | 2 | 1
  Right Ear, 1000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 1000 Hz, <=20 DB HL: Month 12 | 4 | 5
  Right Ear, 1000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 1000 Hz, 21 - 40 DB HL: Month 12 | 1 | 0
  Right Ear, 2000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 2000 Hz, <=20 DB HL: Month 12 | 3 | 4
  Right Ear, 2000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 2000 Hz, 21 - 40 DB HL: Month 12 | 2 | 0
  Right Ear, 4000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 4000 Hz, <=20 DB HL: Month 12 | 4 | 5
  Right Ear, 4000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 4000 Hz, 21 - 40 DB HL: Month 12 | 1 | 0
  Right Ear, 8000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 8000 Hz, <=20 DB HL: Month 12 | 3 | 4
  Right Ear, 8000 Hz, Missing: Month 12: number analyzed (Participants) | 5 | 5
  Right Ear, 8000 Hz, Missing: Month 12 | 2 | 0
  Left Ear, 500 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 500 Hz, <=20 DB HL: Month 12 | 3 | 3
  Left Ear, 500 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 500 Hz, 21 - 40 DB HL: Month 12 | 2 | 1
  Left Ear, 1000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 1000 Hz, <=20 DB HL: Month 12 | 3 | 5
  Left Ear, 1000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 1000 Hz, 21 - 40 DB HL: Month 12 | 2 | 0
  Left Ear, 2000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 2000 Hz, <=20 DB HL: Month 12 | 3 | 4
  Left Ear, 2000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 2000 Hz, 21 - 40 DB HL: Month 12 | 2 | 0
  Left Ear, 4000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 4000 Hz, <=20 DB HL: Month 12 | 4 | 5
  Left Ear, 4000 Hz, 21 - 40 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 4000 Hz, 21 - 40 DB HL: Month 12 | 1 | 0
  Left Ear, 8000 Hz, <=20 DB HL: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 8000 Hz, <=20 DB HL: Month 12 | 3 | 4
  Left Ear, 8000 Hz, Missing: Month 12: number analyzed (Participants) | 5 | 5
  Left Ear, 8000 Hz, Missing: Month 12 | 2 | 1
  Right Ear, 500 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 500 Hz, <=20 DB HL: Month 24 | 5 | 3
  Right Ear, 500 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 500 Hz, 21-40 DB HL: Month 24 | 2 | 0
  Right Ear, 1000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 1000 Hz, <=20 DB HL: Month 24 | 5 | 2
  Right Ear, 1000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 1000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Right Ear, 2000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 2000 Hz, <=20 DB HL: Month 24 | 6 | 3
  Right Ear, 2000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 2000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Right Ear, 4000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 4000 Hz, <=20 DB HL: Month 24 | 7 | 3
  Right Ear, 8000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 8000 Hz, <=20 DB HL: Month 24 | 4 | 3
  Right Ear, 8000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 8000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Right Ear, 8000 Hz, Missing: Month 24: number analyzed (Participants) | 8 | 4
  Right Ear, 8000 Hz, Missing: Month 24 | 1 | 0
  Left Ear, 500 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 500 Hz, <=20 DB HL: Month 24 | 6 | 3
  Left Ear, 500 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 500 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Left Ear, 1000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 1000 Hz, <=20 DB HL: Month 24 | 4 | 3
  Left Ear, 1000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 1000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Left Ear, 2000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 2000 Hz, <=20 DB HL: Month 24 | 6 | 2
  Left Ear, 2000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 2000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Left Ear, 4000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 4000 Hz, <=20 DB HL: Month 24 | 7 | 4
  Left Ear, 8000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 8000 Hz, <=20 DB HL: Month 24 | 3 | 3
  Left Ear, 8000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 8000 Hz, 21-40 DB HL: Month 24 | 1 | 0
  Left Ear, 8000 Hz, Missing: Month 24: number analyzed (Participants) | 8 | 4
  Left Ear, 8000 Hz, Missing: Month 24 | 1 | 0

25. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Air Conduction Via Soundfield Through Pure Tone Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by air conduction via soundfield through pure tone audiometry test which included participants with hearing loss ranged from <=20 DB HL, 21-40 DB HL, 41-70 DB HL, 71-90 DB HL, >90 DB HL or no response, and missing at frequencies ranged from 500 Hz to 4000 Hz at month 12 and 24. Rows according to air conduction categories at specified time points are reported in this outcome measure, only when there was a non-zero data for at least 1 reporting arm.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 13 | 9
Participants
  500 Hz, <=20 DB HL: Month 12 | 6 | 2
  500 Hz, 21-40 DB HL: Month 12 | 5 | 6
  500 Hz, 71-90 DB HL: Month 12 | 1 | 0
  1000 Hz, <=20 DB HL: Month 12 | 9 | 3
  1000 Hz, 21-40 DB HL: Month 12 | 1 | 5
  1000 Hz, 71-90 DB HL: Month 12 | 1 | 0
  2000 Hz, <=20 DB HL: Month 12 | 7 | 2
  2000 Hz, 21-40 DB HL: Month 12 | 3 | 4
  2000 Hz, Missing: Month 12 | 1 | 0
  4000 Hz, <=20 DB HL: Month 12 | 6 | 4
  4000 Hz, 21-40 DB HL: Month 12 | 4 | 4
  4000 Hz, 71-90 DB HL: Month 12 | 1 | 0
  500 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  500 Hz, <=20 DB HL: Month 24 | 6 | 2
  500 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  500 Hz, 21-40 DB HL: Month 24 | 2 | 5
  1000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  1000 Hz, <=20 DB HL: Month 24 | 6 | 6
  1000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  1000 Hz, 21-40 DB HL: Month 24 | 4 | 3
  2000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  2000 Hz, <=20 DB HL: Month 24 | 6 | 3
  2000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  2000 Hz, 21-40 DB HL: Month 24 | 2 | 4
  4000 Hz, <=20 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  4000 Hz, <=20 DB HL: Month 24 | 5 | 4
  4000 Hz, 21-40 DB HL: Month 24: number analyzed (Participants) | 11 | 9
  4000 Hz, 21-40 DB HL: Month 24 | 4 | 3

26. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Tympanometry Assessment (Peak Pressure) Through Immittance Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by tympanometry assessment through immittance audiometry test which included participants with peak pressure signs (+) and (-) at month 12 and 24. In this outcome measure, data have been reported for right and left ear separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: decapascals
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 9 | 8
decapascals
  Peak Pressure for Sign (+), Right Ear: Month 12: number analyzed (Participants) | 7 | 3
  Peak Pressure for Sign (+), Right Ear: Month 12 | 51.89 (63.024) | 27.33 (26.539)
  Peak Pressure for Sign (+), Left Ear: Month 12: number analyzed (Participants) | 3 | 4
  Peak Pressure for Sign (+), Left Ear: Month 12 | 5.07 (4.900) | 73.75 (28.987)
  Peak Pressure for Sign (+), Right Ear: Month 24: number analyzed (Participants) | 3 | 4
  Peak Pressure for Sign (+), Right Ear: Month 24 | 44.00 (46.130) | 33.50 (44.125)
  Peak Pressure for Sign (+), Left Ear: Month 24: number analyzed (Participants) | 7 | 5
  Peak Pressure for Sign (+), Left Ear: Month 24 | 42.71 (50.112) | 35.00 (46.578)
  Peak Pressure for Sign (-), Right Ear: Month 12: number analyzed (Participants) | 6 | 8
  Peak Pressure for Sign (-), Right Ear: Month 12 | 149.3 (144.34) | 67.75 (57.350)
  Peak Pressure for Sign (-), Left Ear: Month 12: number analyzed (Participants) | 9 | 5
  Peak Pressure for Sign (-), Left Ear: Month 12 | 79.89 (64.367) | 46.80 (46.912)
  Peak Pressure for Sign (-), Right Ear: Month 24: number analyzed (Participants) | 8 | 3
  Peak Pressure for Sign (-), Right Ear: Month 24 | 98.00 (55.685) | 83.67 (107.38)
  Peak Pressure for Sign (-), Left Ear: Month 24: number analyzed (Participants) | 6 | 2
  Peak Pressure for Sign (-), Left Ear: Month 24 | 102.2 (84.781) | 135.0 (70.711)

27. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Tympanometry Assessment (Static Acoustic Admittance) Through Immittance Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by tympanometry assessment through immittance audiometry test which included participants with static acoustic admittance at month 12 and 24. In this outcome measure, data have been reported for right and left ear separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimho
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 9 | 11
millimho
  Right Ear: Month 12 | 0.241 (0.1403) | 0.403 (0.1691)
  Left Ear: Month 12: number analyzed (Participants) | 8 | 9
  Left Ear: Month 12 | 0.364 (0.1513) | 0.330 (0.1595)
  Right Ear: Month 24: number analyzed (Participants) | 6 | 6
  Right Ear: Month 24 | 0.273 (0.0784) | 0.400 (0.1321)
  Left Ear: Month 24: number analyzed (Participants) | 8 | 6
  Left Ear: Month 24 | 0.295 (0.0691) | 0.585 (0.5558)

28. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Ipsilateral Stapedial Reflex Through Immittance Audiometry Test
Description: Audiological evaluations of participants were recorded and reported by ipsilateral stapedial reflex through immittance audiometry test which included participants with presence of ipsilateral stapedial reflex at frequencies ranged from 500 Hz to 2000 Hz at month 12 and 24. Ipsilateral stapedial reflex measures are used to assess the neural pathway surrounding the stapedial reflex, which occurs in response to a loud sound (70 to 90 decibel above threshold). In this outcome measure, data have been reported for right and left ear separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 14 | 12
Participants
  500 Hz, Right Ear: Month 12 | 5 | 1
  500 Hz, Left Ear: Month 12 | 6 | 1
  1000 Hz, Right Ear: Month 12 | 5 | 1
  1000 Hz, Left Ear: Month 12 | 6 | 1
  2000 Hz, Right Ear: Month 12 | 5 | 1
  2000 Hz, Left Ear: Month 12 | 6 | 1
  500 Hz, Right Ear: Month 24: number analyzed (Participants) | 13 | 9
  500 Hz, Right Ear: Month 24 | 4 | 2
  500 Hz, Left Ear: Month 24: number analyzed (Participants) | 13 | 9
  500 Hz, Left Ear: Month 24 | 4 | 2
  1000 Hz, Right Ear: Month 24: number analyzed (Participants) | 13 | 9
  1000 Hz, Right Ear: Month 24 | 4 | 2
  1000 Hz, Left Ear: Month 24: number analyzed (Participants) | 13 | 9
  1000 Hz, Left Ear: Month 24 | 5 | 2
  2000 Hz, Right Ear: Month 24: number analyzed (Participants) | 13 | 9
  2000 Hz, Right Ear: Month 24 | 4 | 2
  2000 Hz, Left Ear: Month 24: number analyzed (Participants) | 13 | 9
  2000 Hz, Left Ear: Month 24 | 4 | 2

29. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Transient Evoked Emission Through Otoacoustic Emissions Assessment
Description: Audiological evaluations of participants were recorded and reported by transient evoked emission through otoacoustic emissions assessment which included participants with presence of transient evoked emissions from frequencies 1000 Hz to 4000 Hz at month 12 and 24. In this outcome measure, data have been reported for right and left ear separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 7 | 3
Participants
  1000 Hz, Right Ear: Month 12 | 3 | 2
  1000 Hz, Left Ear: Month 12 | 2 | 1
  1500 Hz, Right Ear: Month 12 | 3 | 2
  1500 Hz, Left Ear: Month 12 | 2 | 2
  2000 Hz, Right Ear: Month 12 | 5 | 2
  2000 Hz, Left Ear: Month 12 | 5 | 2
  3000 Hz, Right Ear: Month 12 | 4 | 2
  3000 Hz, Left Ear: Month 12 | 4 | 2
  4000 Hz, Right Ear: Month 12 | 6 | 2
  4000 Hz, Left Ear: Month 12 | 5 | 3
  1000 Hz, Right Ear: Month 24 | 3 | 2
  1000 Hz, Left Ear: Month 24 | 2 | 2
  1500 Hz, Right Ear: Month 24 | 2 | 3
  1500 Hz, Left Ear: Month 24 | 2 | 3
  2000 Hz, Right Ear: Month 24 | 7 | 3
  2000 Hz, Left Ear: Month 24 | 6 | 3
  3000 Hz, Right Ear: Month 24 | 6 | 3
  3000 Hz, Left Ear: Month 24 | 4 | 3
  4000 Hz, Right Ear: Month 24 | 7 | 3
  4000 Hz, Left Ear: Month 24 | 5 | 3

30. Secondary Outcome: Part B: Audiological Status of Participants as Assessed by Distort Product Through Otoacoustic Emissions Assessment
Description: Audiological evaluations of participants were recorded and reported by distort product through otoacoustic emissions assessment which included participants with presence of distort product at frequencies ranged from 2000 Hz to 8000 Hz at month 12 and 24. Distortion-product otoacoustic emissions (DPOAEs) are generated in the cochlea in response to two tones of a given frequency and sound pressure level presented in the ear canal. Distort product otoacoustic emissions are an objective indicator of normally functioning cochlea outer hair cells. In this outcome measure, data have been reported for right and left ear separately.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 7 | 7
Participants
  2000 Hz, Right Ear: Month 12: number analyzed (Participants) | 6 | 6
  2000 Hz, Right Ear: Month 12 | 4 | 4
  2000 Hz, Left Ear: Month 12: number analyzed (Participants) | 6 | 6
  2000 Hz, Left Ear: Month 12 | 5 | 3
  3000 Hz, Right Ear: Month 12: number analyzed (Participants) | 6 | 6
  3000 Hz, Right Ear: Month 12 | 5 | 4
  3000 Hz, Left Ear: Month 12: number analyzed (Participants) | 6 | 6
  3000 Hz, Left Ear: Month 12 | 5 | 3
  4000 Hz, Right Ear: Month 12: number analyzed (Participants) | 6 | 6
  4000 Hz, Right Ear: Month 12 | 5 | 4
  4000 Hz, Left Ear: Month 12: number analyzed (Participants) | 6 | 6
  4000 Hz, Left Ear: Month 12 | 5 | 3
  6000 Hz, Right Ear: Month 12: number analyzed (Participants) | 6 | 6
  6000 Hz, Right Ear: Month 12 | 4 | 4
  6000 Hz, Left Ear: Month 12: number analyzed (Participants) | 6 | 6
  6000 Hz, Left Ear: Month 12 | 5 | 4
  8000 Hz, Right Ear: Month 12: number analyzed (Participants) | 6 | 6
  8000 Hz, Right Ear: Month 12 | 4 | 2
  8000 Hz, Left Ear: Month 12: number analyzed (Participants) | 6 | 6
  8000 Hz, Left Ear: Month 12 | 5 | 2
  2000 Hz, Right Ear: Month 24 | 4 | 7
  2000 Hz, Left Ear: Month 24 | 4 | 6
  3000 Hz, Right Ear: Month 24 | 7 | 5
  3000 Hz, Left Ear: Month 24 | 6 | 5
  4000 Hz, Right Ear: Month 24 | 6 | 5
  4000 Hz, Left Ear: Month 24 | 6 | 5
  6000 Hz, Right Ear: Month 24 | 4 | 6
  6000 Hz, Left Ear: Month 24 | 5 | 6
  8000 Hz, Right Ear: Month 24 | 3 | 2
  8000 Hz, Left Ear: Month 24 | 4 | 2

31. Secondary Outcome: Part B: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Deaths
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/ incapacity; congenital anomaly. AEs included both serious and all non-serious AEs.
Time Frame: up to 24 months after end of study treatment in Part A (maximum up to 26 months)
Population: Part B safety analysis set included all participants enrolled in Part B of the study for data analyses on developmental progress, audiological, neurological and ophthalmological assessment, and safety.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 27 | 26
Participants
  AEs | 17 | 17
  SAEs | 9 | 6
  Deaths | 0 | 2

32. Secondary Outcome: Part B: Neurological Progress of Participants as Assessed by the Neurology Optimality Score
Description: The Hammersmith Infant Neurological Examination (HINE) was a standard scoring examination to assess development of cranial nerve; posture; movement; tone; and reflexes and reaction. HINE exam global score is a sum of subset (cranial nerve, posture, movement, tone, reflexes and reactions) scores, ranged from 0 to 78, where higher score represents better outcome. Here, the HINE global scores were reported at month 12 and 24.
Time Frame: Month 12 and 24 after end of study treatment in Part A (Day 1 to 14)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Sildenafil | Placebo
Number analyzed (Participants) | 21 | 12
units on a scale
  Neurological Exam Global Score: Month 12 | 69.9 (14.97) | 75.6 (3.45)
  Neurological Exam Global Score: Month 24: number analyzed (Participants) | 17 | 10
  Neurological Exam Global Score: Month 24 | 65.6 (19.71) | 76.5 (2.42)

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to 31 days after end of study drug infusion (up to 45 days); Part B: up to 24 months after end of study treatment in Part A (maximum up to 26 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Groups:
- Part A: IV Sildenafil: Part A: Participants received sildenafil intravenously based on their body weight at a loading dose of 0.1 milligrams per kg (mg/kg) for 30 minutes on Day 1 followed by a maintenance dose of 0.03 milligrams per kg per hour (mg/kg/hr), for a minimum of 2 days and maximum of 14 days. Infusion continuation was upon investigator discretion in view of participants' safety and well-being. Part B: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
- Part A: Placebo: Participants received placebo (0.9 % normal saline or dextrose 10%) at a rate matched to sildenafil infusion, intravenously, based on participant's weight, for a minimum of 2 days and maximum of 14 days. Infusion continuation was upon investigator discretion in view of participants' safety and well-being. Part B: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
- Part B: IV Sildenafil: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
- Part B: Placebo: Part B: Participants who started Part A (not necessarily completed Part A) and who were eligible and consented, continued to be followed up in part B of the study.
Arm/Group | Part A: IV Sildenafil | Part A: Placebo | Part B: IV Sildenafil | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 2/29 | 1/30 | 0/27 | 2/26
Serious Adverse Events (participants affected / at risk) | 7/29 | 2/30 | 9/27 | 6/26
Other Adverse Events (participants affected / at risk) | 20/29 | 19/30 | 14/27 | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: IV Sildenafil (N=29) | Part A: Placebo (N=30) | Part B: IV Sildenafil (N=27) | Part B: Placebo (N=26)
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 1 | 0
Pulmonary malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastroesophageal Reflux (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Congenital heart disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: IV Sildenafil (N=29) | Part A: Placebo (N=30) | Part B: IV Sildenafil (N=27) | Part B: Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 3 | 1 | 0 | 0
Bradycardia neonatal (Cardiac disorders) | 1 | 0 | 1 | 0
Junctional ectopic tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Persistent foetal circulation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Eye oedema (Eye disorders) | 2 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0
Pupil fixed (Eye disorders) | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 4 | 0 | 0 | 0
Drug withdrawal syndrome neonatal (General disorders) | 1 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 3 | 0 | 0
Secretion discharge (General disorders) | 0 | 1 | 0 | 1
Withdrawal syndrome (General disorders) | 0 | 1 | 0 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 1 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 3 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Nosocomial infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Blood albumin decreased (Investigations) | 1 | 0 | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 1
Blood methaemoglobin present (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 2
C-reactive protein increased (Investigations) | 0 | 3 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0
PCO2 decreased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 1 | 0 | 0
Thyroid function test abnormal (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 0 | 1 | 0 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Selective eating disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Haemodynamic instability (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 7 | 3 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Conductive deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypermetropia (Eye disorders) | 0 | 0 | 1 | 1
Strabismus (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 2
Ear infection (Infections and infestations) | 0 | 0 | 4 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 2 | 1
Roseola (Infections and infestations) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Post procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Adenovirus test positive (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood pyruvic acid increased (Investigations) | 0 | 0 | 1 | 0
Gastric residual assessment (Investigations) | 0 | 0 | 0 | 1
Haemoglobin abnormal (Investigations) | 0 | 0 | 0 | 1
Heart rate decreased (Investigations) | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Intra-abdominal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Phrenic nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Psychomotor skills impaired (Nervous system disorders) | 0 | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (3):
  • Study Protocol (2015-04-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT01720524/Prot_000.pdf
  • Statistical Analysis Plan: Redacted SAP Part A of study (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT01720524/SAP_001.pdf
  • Statistical Analysis Plan: Redacted SAP Part B of Study (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT01720524/SAP_002.pdf